CLINICAL TRIAL: NCT06282575
Title: An Open-label Randomized Trial of the Efficacy and Safety of Zanidatamab With Standard-of-care Therapy Against Standard-of-care Therapy Alone for Advanced HER2-positive Biliary Tract Cancer
Brief Title: Efficacy and Safety of Zanidatamab With Standard-of-care Therapy Against Standard-of-care Therapy for Advanced HER2-positive Biliary Tract Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZP598-302; 2023-508219-21-00 (Other: CTIS)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer
Keywords: JZP598; ZW25; HER-2 positive BIliary Tract cancer; Gallbladder Cancer; Intrahepatic Cholangiocarcinoma (ICC); Extrahepatic Cholangiocarcinoma (ECC); Zanidatamab; HER-2 overexpression; HER-2 amplification
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma | interventions — zanidatamab; Cisplatin; Gemcitabine; pembrolizumab; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zanidatamab with Standard-of-care Therapy Arm (Experimental): Zanidatamab plus standard of care treatment of CisGem with or without a PD-1/L1 inhibitor. PD-1/L1 inhibitor will be physician's choice of either Durvalumab or Pembrolizumab, where approved under local regulations.
  Interventions: Drug: Zanidatamab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pembrolizumab; Drug: Durvalumab
- Standard-of-care Therapy Arm (Active Comparator): Standard of care treatment of CisGem with or without a PD-1/L1 inhibitor. PD-1/L1 inhibitor will be physician's choice of either Durvalumab or Pembrolizumab, where approved under local regulations.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Pembrolizumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Zanidatamab — Administered intravenously (IV)
  Other Names: ZW25; JZP598; ZIIHERA®
  Arms: Zanidatamab with Standard-of-care Therapy Arm
Drug: Cisplatin — Administered intravenously (IV)
Drug: Gemcitabine — Administered intravenously (IV)
Drug: Pembrolizumab — Administered intravenously (IV)
Drug: Durvalumab — Administered intravenously (IV)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Zanidatamab plus CisGem (Cisplatin and Gemcitabine) with or without the addition of a programmed death protein 1/ligand-1 (PD-1/L1) inhibitor (physician's choice of either Durvalumab or Pembrolizumab, where approved under local regulations) as first line of treatment for participants with human epidermal growth factor receptor 2 (HER2)-positive biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria

1. Histologically- or cytologically-confirmed Biliary Tract Cancer (BTC), including Gallbladder Cancer (GBC), Intrahepatic Cholangiocarcinoma (ICC), or Extrahepatic Cholangiocarcinoma (ECC).
2. Locally advanced unresectable or metastatic BTC and not eligible for curative resection, transplantation, or ablative therapies.
3. Received no more than 2 cycles of systemic therapy which is limited to Cisplatin and Gemcitabine (CisGem) with or without a PD-1/L1 inhibitor (physician's choice of durvalumab or pembrolizumab, where approved under local regulations) for advanced unresectable or metastatic disease.
4. HER2-positive disease (defined as IHC 3+; or IHC 2+/ ISH+) by IHC and in situ Hybridization (ISH) assay (in participants with IHC 2+ tumors) at a central laboratory on new biopsy tissue or archival tissue from the most recent biopsy.
5. Assessable (measurable or non-measurable) disease as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), per investigator assessment.
6. Male or female ≥ 18 years or age (or the legal age of adulthood per country-specific regulations).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Adequate organ function
9. Females of childbearing potential must have a negative pregnancy test result.
10. Females of childbearing potential and males with a partner of childbearing potential must be willing to use 2 methods of birth control.

Exclusion Criteria

1. Prior treatment with a HER2-targeted agent
2. Prior treatment with checkpoint inhibitors, other than durvalumab or pembrolizumab
3. The following BTC histologic subtypes are excluded: small cell cancer, neuroendocrine tumors, lymphoma, sarcoma, mixed tumor histology, and mucinous cystic neoplasms detected in the biliary tract region.
4. Use of systemic corticosteroids.
5. Brain metastases
6. Severe chronic or active infections
7. History of allogeneic organ transplantation.
8. Active or prior autoimmune inflammatory conditions
9. History of interstitial lung disease or non-infectious pneumonitis.
10. Participation in another clinical trial with an investigational medicinal product within the last 3 months.
11. Females who are breastfeeding
12. Any other medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures.
13. Use of phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in participants with Immunohistochemistry (IHC) 3+ tumors | Up to 52 months
  PFS is defined as the time from the date of randomization to the date of documented disease progression, or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) in participants with IHC 3+ tumors | Up to 68 months
  OS is defined as the time from randomization to death, due to any cause.
Progression Free Survival for all participants | Up to 68 months
  PFS is defined as the time from the date of randomization to the date of documented disease progression, or death from any cause.
OS for all participants | Up to 68 months
  OS is defined as the time from randomization to death, due to any cause.
Number of participants achieving Confirmed objective response rate (cORR) | Up to 68 months
  Confirmed objective response rate is defined as achieving a confirmed best overall response of Complete Response (CR) or Partial Response (PR)
Duration of response (DOR) | Up to 68 months
  Duration of response is defined as the time from the first objective response (CR or PR) to documented Progressive Disease (PD) or death, from any cause.
Number of Patients reporting Treatment-Emergent Adverse Events (TEAE) | Up to 68 months
Maximum serum concentration of Zanidatamab | Up to 68 months
Number of participants who develop Anti-drug antibodies (ADAs) to Zanidatamab | Up to 68 months
Time to definitive deterioration (TDD) for participants with IHC 3+ tumors in patient-reported Physical Functioning (PF) domain score as measured by the EORTC QLQ-C30 | Up to 68 months
  TDD is defined as the time from randomization to the first confirmed clinical meaningful deterioration or death. European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30) final scores range from 0 to 100, where higher scores reflect better functioning
TDD for all participants in patient-reported PF domain score as measured by the EORTC QLQ-C30 | Up to 68 months
  TDD is defined as the time from randomization to the first confirmed clinical meaningful deterioration or death. EORTC QLQ-C30 final scores range from 0 to 100, where higher scores reflect better functioning.
TDD for participants with IHC 3+ tumors in patient-reported symptoms scores as measured by the EORTC QLQ-BIL21 (Pain, Jaundice, Abdominal Pain and Pruritis) | Up to 68 months
  TDD is defined as the time from randomization to the first confirmed clinical meaningful deterioration or death. EORTC Quality of Life Questionnaire - Cholangiocarcinoma and Gallbladder Cancer module (QLQ-BIL21) (Pain, Jaundice, Abdominal Pain, and Pruritis) final scores range from 0 to 100, where higher scores reflect better functioning.
TDD for all participants in patient-reported symptoms scores as measured by the EORTC QLQ-BIL21 (Pain, Jaundice, Abdominal Pain, and Pruritis) | Up to 68 months
  TDD is defined as the time from randomization to the first confirmed clinical meaningful deterioration or death. EORTC QLQ-BIL21 (Pain, Jaundice, Abdominal Pain, and Pruritis) final scores range from 0 to 100, where higher scores reflect better functioning.

CONTACTS AND LOCATIONS:
Locations (183):
- United States (20):
  - City of Hope(City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - AdventHealth Hematology and Oncology, Orlando, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Norton Cancer Institute - Audubon, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Maple Grove, Minnesota
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone - Ambulatory Care Center, New York, New York
  - Memorial Sloan Kettering Cancer Centers, New York, New York
  - Saint Francis Cancer Center, Greenville, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - DFW, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Univerrsity of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University, VCU Health, Richmond, Virginia
- Argentina (8):
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires (caba), Buenos Altes
  - Fundación ARS Médica, San Salvador de Jujuy, Jujuy Province
  - Centro de Investigaciónes Clínicas - Clínica Viedma, Viedma, Río Negro Province
  - Hospital Provincial Del Centenario, Rosario, Santa Fe Province
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario, Santa Fe Province
  - CAIPO Centro para la Atención Integral del Paciente Oncológico, San Miguel de Tucumán, Tucumán Province
  - Centro Médico en Oncología Clínica EXELSUS S.R.L, San Miguel de Tucumán, Tucumán Province
  - Centro Médico Privado CEMAIC, Córdoba
- Belgium (3):
  - Imelda VZW, Bonheiden, Antwerpen
  - UZ Antwerpen, Edegem, Antwerpen
  - UZ Leuven, Leuven, Vlaams-Brabant
- Brazil (8):
  - Liga Norte Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre, Rio Grande do Sul
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre - ISCMPA, Porto Alegrev, Rio Grande do Sul
  - Fundação Pio XII Hospital de Amor de Barretos, Barretos, São Paulo
  - Fundação Doutor Amaral Carvalho - Hospital Amaral Carvalho, Jaú, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto (FUNFARME), São José do Rio Preto, São Paulo
  - Hospital Nossa Senhora Da Conceição/Centro Integrado de Pesquisa em Oncologia CIPO-GHC, Porto Alegre
  - Instituto Nacional de Cancer - INCA, Rio de Janeiro
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Chile (8):
  - Servicios Médicos URUMED SpA, Rancagua, Libertador Gen Bernardo O Higgins
  - Clinica Puerto Montt, Port Montt, Los Lagos Region
  - James Lind Centro de Investigacion del Cancer, Temuco, Región de la Araucanía
  - Centro de Investigacion y Especialidades Medicas (CDIEM), Santiago, Santiago Metropolitan
  - Fundación Arturo López Pérez (FALP), Santiago, Santiago Metropolitan
  - Oncovida, Santiago, Santiago Metropolitan
  - Biocinetic Ltda, Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
- China (10):
  - The First Affiliated Hospital of USTC(Anhui Provincial Hospital), Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Zhongshan Hospital Fudan University, Shanghai
- Czechia (3):
  - Fakultní nemocnice Brno, Interní hematologická a onkologická klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Klinika onkologie a radioterapie, Hradec Králové
  - Fakultni nemocnice v Motole, Onkologicka klinika, Prague
- Finland (3):
  - Docrates Cancer Center, Helsinki
  - Comprehensive Cancer Center, Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- France (11):
  - CHU de Toulouse- (Toulouse University Hospital Center), Toulouse, Cedex 9
  - CHU Besancon, Besançon, Cedex
  - CHU de Bordeaux - Hôpital Haut Leveque, Pessac, Cedex
  - CHU Brest Hôpital de la Cavale Blanche, Brest
  - CHU Estaing, Clermont-Ferrand
  - Hospital Beaujon University, Clichy
  - Hopital Henri Mondor, Créteil
  - CHU Montepellier - Hôpital Saint Eloi, Montpellier
  - CHU Poitiers, Poitiers
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (10):
  - Universitätsklinikum Freiburg - Klinik für Innere Medizin II,, Freiburg im Breisgau, Baden-Wurttemberg
  - Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen - Medizinische Universitätsklinik, Innere Medizin I, Tübingen, Baden-Wuttemberg
  - LMU Universitätsklinikum München, Campus Großhadern, Medizinische Klinik und Poliklinik III - Hämatologie und Onkologie, München, Bavaria
  - Krankenhaus Nordwest - Institut für Klinisch-Onkologische Forschung (IFK), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover - Klinik Fur Gastroenterologie, Hepatologie, Infektiologie und Endokrinologie, Hanover, Nieder-Sachsen
  - Technische Universität Dresden Medizinische Fakultät Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Medizinische Klinik I (MKI), Lübeck, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin - Campus Virchow Klinikum, Medizinische Klinik mit Schwerpunkt Hamatologie und Tumorimmunologie, Berlin
  - Asklepios Tumorzentrum Hamburg, Asklepios Klinik Altona - Onkologie und Palliativmedizin mit Sektionen Hamatologie und Rheumatologie, Hamburg
- India (8):
  - KLES Dr Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Chopda Medicare & Research Centre Pvt. Ltd - Magnum Heart Institute, Nashik, Maharashtra
  - AIG Hospitals (A Unit of Asian Institute of Gastroenterology), Hyderabad, Telangana
  - Pi Health Cancer Hospital, Hyderabad, Telangana
  - Mahamana Pandit Madan Mohan Malviya Cancer Centre, Varanasi, Uttar Pradesh
  - Max Super Speciality Hospital - Saket (a unit of Devki Devi foundation), New Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - The Hadassah University Medical Center, Ein Kerem Hospital, Jerusalem
  - Rabin Medical Center, Bellinson Hospital, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Hashomer, Ramat Gan, HaMerkaz
  - Tel Aviv Sourasky Medical Center (Ichilov), Tel Aviv
- Italy (11):
  - Azienda Ospedaliero Universitaria di Cagliari Presidio Ospedaliero Duilio Casula, Monserrato, Cagliari
  - Instituo di Candiolo, Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo, Torino
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Istituto Nazionale per lo studio e la cura dei Tumori, Milan
  - AOU dell'Universit~ degli Studi della Campania Luigi Vanvitelli, Napoli
  - Veneto Institute of Oncology IOV - I.R.C.C.S., Padua
  - Azienda Ospedaliero - Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Gemelli-IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Sanitaria Universitaria Friuli Centrale - P.O. S. Maria della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (20):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyôto
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka, Osaka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Yamaguchi University Hospital, Ube-Shi, Yamaguchi
  - Osaka University Hospital, Suita-Shi, Ôsaka
- Portugal (5):
  - Unidade Local de Saude de Almada-Seixal, E.P.E. - Hospital Garcia de Orta, Almada
  - Unidade Local de Saude de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Unidade Local de Saúde de São José - Hospital de Santo António dos Capuchos, Lisbon
  - Champalimaud Clinical Center, Lisbon
  - Instituto Português de Oncologia Do Porto Francisco Gentil, EPE, Porto
- Hospital Oncologico, Puerto Rico Medical Center, Rio Piedras, Puerto Rico
- Romania (4):
  - Spital Clinic Judetean de Urgenta Bihor, Oradea, Bihor County
  - Centrul De Oncologie "SF. Nectarie" S.R.L., Craiova, Dolj
  - Institutul Clinic Fundeni, Bucharest
  - Centrul de Oncologie Euroclinic SRL, Iași
- Serbia (3):
  - University Clinical Center of Serbia, Clinic for Gastroenterohepatology, Belgrade
  - Military Medical Academy, Clinic for Gastroenterology and Hepatology, Belgrade
  - Oncology Institute of Vojvodina, Internal Oncology Clinic, Kamenitz
- South Korea (11):
  - CHA Bundang Medical Center, CHA University, Bundang-Gu, Seongnam-Si, Gyeonggi-do
  - National Cancer Center, Ilsandong-gu, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (11):
  - Complejo Hospitalario Universitario de Santiago -Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna
  - Vall d'Hebron Institute of Oncology/Hospital Universitari de Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Onkologiska mottagningen, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Cancerstudieenheten Huddinge, Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Onkologiska mottagningen, Skånes Universitetssjukhus Malmö, Malmo
- Taiwan (5):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung Branch of the Chang Gung Medical Foundation, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Cancer Center, Taipei
  - Chang Gung Memorial Hospital Linkou Branch of the Chang Gung Medical Foundation, Taoyuan District
- Turkey (Türkiye) (4):
  - Istanbul University Cerrahpasa Medical Faculty Hospital/Clinical Research Center, Istanbul, Fatih
  - Hacettepe University Cancer Institute, Ankara, Sihhiye
  - Akdeniz University Medical Faculty Hospital, Antalya
  - Trakya University Faculty of Medicine, Edirne
- United Kingdom (5):
  - Mount Vernon Cancer Centre, London, England
  - NHS Foundation Trust Royal Marsden Hospital, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Royal Marsden Hospital NHS Foundation Trust, Surrey, England
  - Western General Hospital, Edinburgh Cancer Centre, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: No